CLINICAL TRIAL: NCT04183855
Title: The Relationship Between Blood Glucose and Satiety Ratings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Principal Investigator, Western University, Canada
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 115099
Record Dates: First submitted 2019-11-26; First posted 2019-12-03 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-11

CONDITIONS: Satiety; Appetite

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Experimental): no supplement will be provided on the day of the experiment
  Interventions: Behavioral: satiety ratings
- Generation UCAN (Experimental): carbohydrates - protein (Generation UCAN supplement, 250ml, 10% solution)
  Interventions: Dietary Supplement: Generation UCAN supplementation; Behavioral: satiety ratings
- Mirexus PhytoSpherix (Experimental): carbohydrates alone (Mirexus PhytoSpherix, 250ml, 10% solution)
  Interventions: Dietary Supplement: Mirexus PhytoSpherix supplementation; Behavioral: satiety ratings

INTERVENTIONS:
Dietary Supplement: Generation UCAN supplementation — carbohydrates - protein (Generation UCAN supplement, 250ml, 10% solution)
  Arms: Generation UCAN
Dietary Supplement: Mirexus PhytoSpherix supplementation — carbohydrates alone (Mirexus PhytoSpherix, 250ml, 10% solution)
  Arms: Mirexus PhytoSpherix
Behavioral: satiety ratings — questionnaire on satiety ratings will be provided to participants 15, 30, 45 and 60 min after the drink (or no drink)

SUMMARY:
Participants will be given a drink (and no drink for one of the treatments) prior to a pizza dinner. Ratings on satiety, appetite and desire to eat will be asked with the use of a questionnaire. Blood glucose will also be measured. One hour after the drink, participants will be given a pizza and can eat as much as they want. The pizza remaining will be weighed.

DETAILED DESCRIPTION:
Each participant will receive all three treatments on separate occasions in random order (separated by a week). The three treatments include control (no supplement), carbohydrates - protein (Generation UCAN supplement, 250ml, 10% solution) and carbohydrates alone (Mirexus PhytoSpherix, 250ml, 10% solution). Participants will report to the lab between 4-5 pm and 4 hours after their last meal on day they have not exercised. Participants will record food intake the day of the first experiment and will be asked to replicate both type and quantity for subsequent visits. Upon arrival at the lab, baseline measures (blood glucose as well as rating of satiety ratings, appetite and desire to eat (10-point visual analogue scale). Then the treatment will be given and all the aforementioned variables will be remeasured at 15, 30, 45 and 60 minutes post drink. At 65 minutes, participants will be provided with an ad libitum pizza meal. Participants will be told to eat until they are "comfortably full" (Bellissimo et al., 2008). The pizza provided will be weighed initially and once the participant is done eating and has left the lab, the remaining pizza will be weighed and recorded. The pizza will be a cheese only pizza to minimize any difference in energy intake due to the location of additional items placed on the pizza.

Participants will not be told the true purpose of this experiment, instead they will be told that the pizza meal is a reward for participating in the study. Later, at the conclusion of the study all will be debriefed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females at the age of 18-40
* sedentary individuals

Exclusion Criteria:

* exercise more than twice per week
* does not like pizza
* do not eat three meals a day
* medications that affect eating patterns
* have metabolic and gastrointestinal diseases

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
changes in satiety ratings after the drink | 15, 30, 45, 60 min after the drink
  satiety ratings will be asked with the use a 10 point visual analog scale (VAS) questionnaire, 10 being do not want to consume any more food and 1 being strong desire to consume food
Food intake | 90 min after the drink
  food intake after each treatment will be measured by weighing the left over pizza slices

SECONDARY OUTCOMES:
changes in appetite ratings after the drink | 15, 30, 45, 60 min after the drink
  appetite ratings will be asked with the use a 10 point visual analog scale (VAS), 10 being strong desire to consume food and 1 being no desire to consume food at all
changes in blood glucose after the drink | 15, 30, 45, 60 min after the drink
  blood glucose will be measured through finger pricks
changes in desire to eat ratings | 15, 30, 45, 60 min after the drink
  desire to eat ratings will be asked with the use a 10 point visual analog scale (VAS), 10 being no desire to eat at all and 1 being strong desire to eat

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PhD, Principal Investigator — Western University
Locations (1):
- Exercise Nutrition Laboratory (Western University), London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No